CLINICAL TRIAL: NCT02830399
Title: Clinical Trial on Efficacy of Repeated Transcranial Magnetic Stimulation (rTMS) to Improve Electroconvulsive Therapy (ECT) in Treatment-Resistant Depression (TRD): STIMAGNECT Study
Brief Title: Clinical Trial on Efficacy of rTMS to Improve ECT in Treatment-Resistant Depression
Acronym: STIMAGNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier du Rouvray (Other Government)
Collaborators: University Hospital, Rouen (Other); Centre Hospitalier Henri Laborit (Other); University Hospital, Caen (Other)
Responsible Party: Principal Investigator, Maud Rothärmel, M.D., Centre Hospitalier du Rouvray
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-A01810-49
Record Dates: First submitted 2016-06-08; First posted 2016-07-12 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Major Depressive Disorder
Keywords: treatment-resistant-depression; rTMS; ECT; Augmentation strategy
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- active rTMS-ECT (Active Comparator): 5 active high frequency rTMS before 5 bilateral ECT
  Interventions: Device: active rTMS-ECT
- sham rTMS-ECT (Placebo Comparator): 5 sham rTMS before 5 bilateral ECT
  Interventions: Device: sham rTMS-ECT

INTERVENTIONS:
Device: active rTMS-ECT — 5 High Frequency (20Hz) rTMS (applicated on the left prefrontal dorsolateral cortex) before 5 bilateral ECT
  Arms: active rTMS-ECT
Device: sham rTMS-ECT — 5 sham rTMS (applicated on the left prefrontal dorsolateral cortex) before 5 bilateral ECT
  Arms: sham rTMS-ECT

SUMMARY:
It's a prospective, multicentric, randomized, controlled study concerning 56 patients with treatment-resistant depression (TRD). The main objective of this study was to evaluate the efficacy of priming repeated Transcranial Magnetic Stimulation (rTMS) sessions before Electroconvulsive therapy (ECT) for treatment of TRD patients. The primary outcome will be the depressive symptoms intensity measured with the Hamilton Rating Scale For Depression (HAMD-21 items) after 5 ECT. The secondary outcome is to evaluate the safety and most particularly the cognitive effects of this association.

DETAILED DESCRIPTION:
Included patients are adults, aged between 18 and 70 years, with major depression (Hamilton Rating scale for Depression, HAMD ≥ 15). Patients don't have any experience concerning repeated Transcranial Magnetic Stimulation (rTMS).

Patients with treatment-resistant depression (TRD) were assigned to two treatment groups in addition to their current pharmacotherapy regimen : one group received 5 active-rTMS before Electroconvulsive therapy (ECT) and the other one received sham-rTMS before ECT. The depressive symptoms and the cognitive functions are evaluated before rTMS, after 5 rTMS and after 5 ECT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Major Depressive Disorder (HAMD≥15)
* Level of resistance ≥ 3 (Thase and Rush)
* Participants who gave their informed, written consent

Exclusion Criteria:

* Contraindication of Electroconvulsive therapy (ECT), repeated Transcranial Magnetic Stimulation (rTMS), Magnetic Resonance Imaging (MRI), anesthesia
* History of epilepsy; severe neurological or systemic disorder that could significantly affect cognition
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Relative improvement of the Hamilton Rating Scale for Depression 21-items score | Relative improvement of the Hamilton Rating Scale for Depression score between the inclusion and 19 days after the inclusion

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Centre Esquirol- CHU de Caen, Caen
  - Centre Hospitalier Laborit, Poitiers
  - Centre Hospitalier du Rouvray, Sotteville-lès-Rouen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rotharmel M, Quesada P, Husson T, Harika-Germaneau G, Nathou C, Guehl J, Dalmont M, Opolczynski G, Mirea-Grivel I, Millet B, Gerardin E, Compere V, Dollfus S, Jaafari N, Benichou J, Thill C, Guillin O, Moulier V. The priming effect of repetitive transcranial magnetic stimulation on clinical response to electroconvulsive therapy in treatment-resistant depression: a randomized, double-blind, sham-controlled study. Psychol Med. 2023 Apr;53(5):2060-2071. doi: 10.1017/S0033291721003810. Epub 2021 Sep 28. PMID 34579796